CLINICAL TRIAL: NCT02217111
Title: Prospective Study of Voice Therapy in Children: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kittie Verdolini Abbott, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO14060563
Record Dates: First submitted 2014-07-09; First posted 2014-08-15 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Vocal Fold Nodules
Keywords: vocal fold nodules; pediatric; voice therapy; acoustic; aerodynamic; quality of life; Adventures in Voice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- voice therapy (Experimental)
  Interventions: Behavioral: Adventures in Voice: Pediatric Voice Therapy

INTERVENTIONS:
Behavioral: Adventures in Voice: Pediatric Voice Therapy

SUMMARY:
The purpose of this prospective study is to obtain preliminary data on changes in pre-post voice therapy outcomes in children diagnosed with vocal fold nodules, as a function of a series of cognitive operations. The primary outcome is voice-related quality of life (questionnaire). Secondary outcomes are standard acoustic and aerodynamic measures derived from sustained vowel and running speech samples.

DETAILED DESCRIPTION:
* Voice disorders are the most common communication disorder across the lifespan, affecting more than 5 million school-aged children annually in the United States.
* Vocal fold nodules are the most frequent pathology affecting voice in children, and may affect up to 21% of the pediatric population at any given point in time.
* Children with voice disorders caused by this and other conditions often experience negative consequences in quality of life and academic participation.
* Specifically, these children are at increased risk for inferior school performance, dysfunctional psychosocial development, and other negative sequelae.
* Overwhelmingly, the first-line treatment for voice problems due to nodules is behavioral voice therapy.
* Unfortunately, the pediatric population is badly underserved by Speech-Language Pathology for this condition and others affecting voice.
* Moreover, to date, experimental findings on the benefits of voice therapy in children have not been reported.
* In the present study, children who present with voice complaints to the Department of Otolaryngology at Children's Hospital of Pittsburgh (CHP), who are diagnosed with vocal fold nodules, and who following informed consent are found to satisfy other inclusion criteria detailed shortly, will be eligible for participation in the study.
* Eligible children will undergo a 45-60-min battery of standardized tests evaluating simple cognitive functions.
* Participation in the protocol will not depend on the outcome of these tests.
* Then, all children will receive an increasingly used, 9-week program of voice therapy for children with vocal fold nodules and other conditions affecting voice, "Adventures in Voice," a program grounded in basic biomechanical, biological, and cognitive science.
* Dependent variables will be pre- to post-therapy change in voice-related quality-of-life, based on the Pediatric Voice-Related Quality of Life Survey (Boseley, Cunningham, Volk, & Hartnick, 2006) (primary outcome measure) and change in a series of standard acoustic and aerodynamic measures based on sustained vowel and simple running speech samples, described shortly (secondary outcome measures).
* The independent variables involve a series of cognitive measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of vocal fold nodules.
* Age 4-11 yr.
* Informed Consent.
* English comprehension and production sufficient to participate in the protocol and in voice therapy.
* Considered behaviorally and cognitively appropriate by the ear, nose, and throat physician and speech-language pathologist for voice therapy.
* Parent and child willingness to participate in all aspects of the protocol and voice therapy.

Exclusion Criteria:

* Co-morbid medical conditions or medications that would mask or amplify the outcome of voice therapy, including (a) developmental or other neuromuscular conditions, (b) major illness, chronic or acute, with the exception of laryngopharyngeal reflux disease (LPR) or allergies and their treatments, which are common in both children and adults with voice disorders, thus their exclusion would severely restrict the participant pool and, moreover, threaten external validity.
* Hearing loss: > 20 dB hearing loss at 1000, 2000, 4000 Hz in at least one ear.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pediatric Voice-Related Quality of Life Survey (PVRQOL) | 13-16 weeks
  The PVRQOL is a 10-item instrument designed and validated as a self-administered and parent-proxy-administered instrument for the pediatric population with voice disorders to measure both social-emotional and physical-functional aspects of voice problems. The PVRQOL raw scores are transformed to a scale of 0-100 for easy of interpretation. The PVRQOL will be administered prior to initiation of voice therapy as well as one week post-voice therapy termination.

SECONDARY OUTCOMES:
Spectral and Cepstral Analysis | 13-16 weeks
  Cepstral peak measures and associated Spectral measurements will be obtained using the Analysis of Dysphonia in Speech and Voice (ADSV) program for the following voice sample tasks: (1) sustained vowel /a/, (2) standard sentences (based on the Consensus Auditory-Perceptual Evaluation of Voice, 2006), and (3) counting from 1-10. The ADSV program will provide the following seven (7) key measures obtained from Spectral, Cepstral, or combination of Spectral and Cepstral measures: (1) The Cepstral Peak Prominence (CPP), (2) The Cepstral Peak Prominence standard deviation (CPP sd); (3) The Low/High Spectral Ratio (L/H Ratio using a default cutoff of 4 kHz); (4) The L/H Ratio standard deviation; (5) The CPP frequency (an estimate of the fundamental frequency (F0) obtained form the Cepstral peak); (6) The CPP frequency standard deviation; and (7) The Cepstral Spectral Index of Dysphonia (CSID) - a multivariate acoustic estimate of dysphonia severity using a 100mm visual analog scale (VAS).
Vital Capacity (Aerodynamic Analysis) | 13-16 weeks
  Hand held spirometry (EasyOne) will be used to obtain estimates of Vital Capacity. The Vital Capacity measure will be used to calculate estimated laryngeal airflow with phonatory quotient (VC (mL/s) / MPT (s)).These measures will be performed at baseline and one-week post-therapy follow up.
Developmental Neuropsychological Assessment (NEPSY) (Cognitive Assessment) | 13-16 weeks
  This test evaluates executive function, memory, attention, and sensorimotor functions, and is completed by the child. It is standardized for children ages 3-16 yr. The test will be administered before pre- and post- voice therapy.
Browns ADD Scales (Cognitive Assessment) | 13-16 weeks
  These Scales evaluate potential Attention Deficit Disorder (ADD), but may be appropriate for children without ADD as well. This test is completed by the guardian, and can be administered concurrently with administration of other tests to the child. The battery will be administered pre- and post-voice therapy.
Children's Memory Scale (Cognitive Assessment) | 13-16 weeks
  This test assesses verbal and visual short- and long-term memory. It is standardized for children as young as 5 yr of age, but most 4-yr-old children should be able to complete the test. The test will be administered before pre- and post- voice therapy.
Maximum Phonation Time (Aerodynamic Analysis) | 13-16 weeks
  Will provide indirect estimates of respiratory, in relation to phonatory, function. These measures will be performed at baseline and one-week post-therapy follow up.
S/Z Ratio (Aerodynamic Analysis) | 13-16 weeks
  Will provide indirect estimates of respiratory, in relation to phonatory, function. These measures will be performed at baseline and one-week post-therapy follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Verdolini Abbott, Ph.D., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania